CLINICAL TRIAL: NCT04063436
Title: Evaluation of a New Nasal Pillows Mask for the Treatment of Obstructive Sleep Apnea
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Clinical trial was cancelled
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-264
Record Dates: First submitted 2019-08-13; First posted 2019-08-21 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: After the baseline period, all participants will be trialed on the same new nasal pillows mask.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Experimental (Experimental): Participants will be placed in the experimental arm for 14±5 days, during which they will be using the new nasal pillows mask for PAP therapy.
  Interventions: Device: New nasal pillows mask with PAP therapy

INTERVENTIONS:
Device: New nasal pillows mask with PAP therapy — Participants will be placed in the experimental arm for 14±5 days, during which they will be using the new nasal pillows mask for PAP therapy.

SUMMARY:
This clinical trial is designed to evaluate the performance, comfort, and usability of a new nasal pillows mask for the treatment of obstructive sleep apnea (OSA) in a home environment.

ELIGIBILITY:
Inclusion Criteria:

* Are ≥22 years of age
* Weigh ≥66 lbs
* Have been formally diagnosed with OSA by a physician
* Have an AHI ≥5 on a diagnostic night
* Have been prescribed PAP therapy to treat OSA by a physician
* Are an existing nasal pillows mask user
* Have been using a nasal pillows mask for ≥3 months prior to enrolment into the study
* Are compliant with PAP therapy for ≥4 hours per night for 70% of nights
* Are fluent in spoken and written English
* Possess the capacity to provide informed consent

Exclusion Criteria:

* Are intolerant to PAP therapy
* Possess, or suffer from, anatomical or physiological conditions which make PAP therapy inappropriate
* Are currently diagnosed with respiratory disease or CO2 retention
* Are pregnant or think they may be pregnant
* Have an IPAP pressure of >25 cmH2O
* Persons who use a PAP therapy machine for the delivery of medicines, except O2
* Use a PAP therapy machine that does not possess data recording capabilities to capture AHI and leak information that is accessible to OSMI

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-23 (Estimated); Primary Completion 2019-10-11 (Estimated); Study Completion 2019-10-11 (Estimated)

PRIMARY OUTCOMES:
Performance of new nasal pillows mask | 14±5 days
  The new nasal pillows mask provides adequate PAP therapy for OSA when used in a home environment. This is an objective measure and is determined by the Apnea-Hypopnea Index recorded on PAP therapy machines.

SECONDARY OUTCOMES:
Comfort of new nasal pillows mask | 14±5 days
  The new nasal pillows mask is comfortable during PAP therapy for OSA when used in a home environment. This is a subjective measure and is determined by a five-point Likert-type scale as recorded on a questionnaire.
Usability of new nasal pillows mask | 14±5 days
  The new nasal pillows mask is user-friendly during PAP therapy for OSA when used in a home environment. This is a subjective measure and is determined by a five-point Likert-type scale as recorded on a questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio Sleep Medicine Institute, Dublin, Ohio, United States

IPD SHARING:
Plan to Share IPD: No